CLINICAL TRIAL: NCT03701022
Title: An Open-lable, Single Arm, Single Center, Phase 2 Study of PD1 Combined With Apatinib in Patients With Relapsed or Refractory NK/T Cell
Brief Title: PD1 Combined With Apatinib in Patients With Relapsed or Refractory NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Party secretary of Cancer Hospital of Peking University，Director of Internal Medicine, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-APTN-IIT-NKT lymphoma
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR1210 +Apatinib (Experimental): SHR-1210 injection, 200 mg/dose, intravenous infusion within 20-60 minutes.
  Interventions: Drug: SHR1210

INTERVENTIONS:
Drug: SHR1210 — SHR-1210 injection, 200 mg/dose, intravenous infusion within 20-60 minutes. Apatinib oral administration, 500mg per day.
  Other Names: Apatinib

SUMMARY:
This is an open-label, single-center, nonrandomized, Phase 2 study to evaluate efficacy and safety of SHR-1210 combined with Apatinib in subjects with relapsed or refractory NK/T cell lymphoma.Efficacy will be assessed every 8 weeks according to 2014 Lugano criteria.Safety evaluations (both clinical and laboratory) are performed at baseline, before each study treatment, and throughout the study.

DETAILED DESCRIPTION:
The primary objective of this phase 2 study is to assess objective response rate of SHR-1210 combined with Apatinib in patients with relapsed or refractory NK/T cell lymphoma. The secondary objective is to observe time to response,progression free survival rate at 2 years,overall survival rate at 2 years，safety and immunogenicity of SHR-1210 combined with Apatinib in relapsed or refractory NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed extranodal NK/T cell lymphoma nasal, PTCL,NOS, AITL, ALCL;
2. Subjects must be recurrent or refractory, and 10-15 white tumors of tumor tissue should be provided.
3. Subjects enrolled have measurable lesion(s) according to Lugano 2014 criteria
4. ECOG performance status of 0 or 1;

6.Life expectancy ≥ 12 weeks.; 7.Adequate laboratory parameters during the screening period as evidenced by the following:

a.Absolute neutrophil count ≥ 1.5× 109/L ; b.Platelets ≥ 100 × 109/L; c.Hemoglobin ≥ 9.0 g/dL; d.Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), ALT and AST ≤ 2.5×ULN e.Serum Creatinine ≤1.25×ULN or Creatinine clearance≥45 mL/min; f.Coagulation function index：INR ≤1.5×ULN，APTT≤1.5×ULN 8.Women of childbearing potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 120 days after receiving the last dose of study treatment. Women of childbearing potential with pregnancy test negative within 7days before entering the group and not in in lactation; Male subjects with WOCBP partner should receive Surgical sterilization orconsent to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 120 days after receiving the last dose of study treatment.

9.Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Known central nervous system lymphoma
2. Haemophilus cell syndrome at diagnosis
3. Large lung vessels were involved
4. History and complication

   1. Active, known or suspected autoimmune disease. Subjects who were in a stable state without systemic immunosuppressive therapy were admitted
   2. Subjects requiring systemic treatment with corticosteroids (> 10 mg/day prednisone or equivalent) or other immunosuppressive agents were given the study drug within 14 days prior to administration. Inhaled or topical corticosteroids and adrenaline replacement at a therapeutic dose of more than 10 mg/day prednisone are allowed in the absence of active autoimmune disease
   3. Recieved anti-tumor vaccines or other anti-tumor therapy with immune stimulation within 3 months.
   4. Prior exposure to any PD-1/PD-L1/PD -L 2 or CTLA -4 antibody .
   5. Participating in other clinical studies or less than 4 weeks before the end of a clinical trial;
   6. Known and suspicion of interstitial pneumonia
   7. History of other malignancies except in patients with basal cell carcinoma of the skin, superficial bladder, squamous cell carcinoma of the skin, or carcinoma of the cervix in situ who had undergone potential curable treatment and had no recurrence within five years of initiation of self-treatment;
   8. Received chemotherapy, radiotherapy,immunotherapy, including topical therapy within 4 weeks. Previous anti-tumor therapy related adverse reactions (except trichomadesis) did not recover to CTCAE ≤1.
   9. Prior allo-HSCT.
   10. ASCT within 90 days.
   11. Impact of major surgery or severe trauma had been eliminated for less than 14 days.
   12. Active pulmonary tuberculosis.
   13. Severe acute or chronic infection requiring systemic therapy.
   14. In the first 2 months before treatment, there was a significant amount of half a teaspoon (2.5ml) of blood or hemoptysis
   15. Significant clinical symptoms of bleeding or a clear tendency to bleed occurred within the first three months of randomization, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ or above, or vasculitis, etc;
   16. Arteriovenous thrombotic events, such as cerebral vascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism, occurred within the first six months of treatment.
   17. Known hereditary or acquired bleeding and thrombotic tendencies ;
   18. Suffering from hypertension, and the treatment of hypotensive drugs can not get good control.(systolic blood pressure is greater than 140 mmHg or diastolic pressure is more than 90 mmHg);
   19. Suffering from heart failure (New York Heart Association standard III or IV) and given appropriate medical treatment.Uncontrolled coronary artery disease and arrhythmia. History of myocardial infarction within 6 months;
   20. Live vaccinations were given within four weeks before the study drug was administered. Inactivated viral vaccines for seasonal influenza were allowed, but live attenuated influenza vaccines for intranasal use were not allowed.
5. laboratory test

   1. known HIV positive or known AIDS.
   2. Untreated active hepatitis; Hepatitis B and hepatitis C infection in common.
   3. Abnormal coagulation function (PT > 16s, APTT > 43s, TT > 21s, Fbg < 2G / L) having tends to bleed or is undergoing thrombolytic or anticoagulant therapy;
   4. Routine urine tests indicate that urine protein is more than + +, or 24 hours urine protein is more than 1 g.
6. Other factors that may lead to the study termination, such as severe disease or abnormal laboratory tests or family or social factors affecting subjects safety or test data and sample collection
7. Women suffering from pregnancy or lactation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2020-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate | from first patient first visit to 6 month after last patient first visit
  rate of subjects achieved complete response plus partial response in all evaluable subjects

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, Principal Investigator — Cancer Hospital of Beijing University

IPD SHARING:
Plan to Share IPD: No